CLINICAL TRIAL: NCT05689905
Title: Immunologic Risk of Pregnancy in Women With Lung Transplant
Brief Title: Immunologic Risk of Pregnancy in Women With Lung Transplantion : a National Multicentric Study
Acronym: TRIGGER-2
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: Institut de Recherche en Santé Respiratoire (Unknown)
Responsible Party: Sponsor
Other Study IDs: RC22_0581
Record Dates: First submitted 2022-11-30; First posted 2023-01-19 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Lung Transplantation; Graft Rejection; Pregnancy
Keywords: Lung Transplantations; Pregnancy; Transplant Rejection; Transplantation Immunology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva swab from the mother's child with a lung transplant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Common HLA antigens with the lung donor: Children who have common HLA antigens with the lung donor of their mother
  Interventions: Diagnostic Test: HLA typing of the children
- No common HLA antigens with the lung donor: Children without common HLA antigens with the lung donor of their mother.
  Interventions: Diagnostic Test: HLA typing of the children

INTERVENTIONS:
Diagnostic Test: HLA typing of the children — The HLA typing is made on a mouth swab of the children, that is a painless non-invasive procedure.

SUMMARY:
TRIGGER 1 is a previous study that evaluate the immunological risk of pregnancy in women with lung transplants in France, whose pregnancy has ended between January 1, 2012 and December 31, 2021. The primary endpoint is the occurrence of humoral rejection with a year after pregnancy.

TRIGGER 2 aims to evaluate the risk of humoral rejection if there are common antigens between the child and the lung donor. We will collect HLA typing from children to compare them to the HLA typing of the mother, the lung donor and the antibodies produced if there are.

Thus, it will help us to suggest recommendations to limit the immunological risk of pregnancy for lung transplant women.

Lung transplantation is the treatment of choice of terminal chronic respiratory failure, such as cystic fibrosis and pulmonary hypertension. Young female patient of childbearing age are concerned.

For many years, given the risk of maternal and fetal complications, pregnancies were not recommended. Studies on large cohorts of transplanted patients, particularly kidney transplanted patients, have made it possible to study the risks of maternal, obstetrical and neonatal complications.

A few studies have been published in lung transplantation on small numbers of patients. However, these publications reporting on the fate of pregnancies in cohorts of lung transplant patients do not mentioned the immunological risk, with in particular the absence of studies on the risk of humoral rejection, appearance of anti-HLA (Human Leukocyte Antigens) antibodies (Ac) and the possible appearance of anti-HLA Ac directed against the donor (donor specific antibody, DSA).

TRIGGER 1 is a previous study, whose main objective is to evaluate the immunological risk of pregnancy in women with lung transplants (mono-, bi-, or cardiopulmonary) in France, whose pregnancy has ended between January 1, 2012 and December 31, 2021. The primary endpoint is the occurrence of humoral rejection within 1 year after pregnancy.

For this study TRIGGER2, we will collect the HLA typing of the children for pregnancies that resulted in the birth of a child. Thus, we will be able to compare the HLA typing of the children with the HLA typings of the mother and the lung donor, and the antibodies produced by the mother. The primary endpoint is to evaluate the risk of humoral rejection if there are common HLA antigens between the child and the lung donor.

ELIGIBILITY:
Inclusion Criteria:

* Children born between 01/01/2012 and 31/12/2021 of female patients over 18 years old with lung transplantation (mono, uni or cardio pulmonary) in France,
* Alive at the time of our study.
* Legal guardians' consent for oral swabbing of their child and HLA typing on this swab
* Affiliated or beneficiaries of a social security system or similar

Exclusion Criteria:

- Refusal of consent by the patient and/or one of the two parents

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Cohort of female lung transplant patients, a rare pathology, and their children.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Risk of humoral rejection if common HLA antigen between child and graft. | Baseline
  Identification of common HLA antigen between child and graft by HLA typing

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - Nantes University Hospital, Nantes, Loire Atlantique
  - Bordeaux University Hospital, Bordeaux
  - Grenoble University Hospital, Grenoble
  - Marie Lannelongue Hospital (GHSJ), Le Plessis-Robinson
  - Civils Hospitals Lyon, Lyon
  - AP-HM, Marseille
  - Cochin Hospital (AP-HP), Paris
  - Strasbourg University Hospital, Strasbourg
  - Foch Hospital, Suresnes

IPD SHARING:
Plan to Share IPD: No